CLINICAL TRIAL: NCT01894945
Title: Dual Time Point PET in Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Karen Juul Mylam, MD, Odense University Hospital
Other Study IDs: 10.06b
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Hodgkin's and Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with suspected lymphoma.

SUMMARY:
This study aims to investigate the value of dual time point PET/CT in lymphoma. Since FDG uptake is linked to glucose metabolism, PET imaging is also used to detect suspected sites for infectious and inflammatory disorders. In a clinical setting, it is a challenge to distinguish between FDG uptake in benign and malignant lesions and this gives rise to a considerable quantity of false positive results and decreased positive predictive values. Performing FDG-PET imaging sixty minutes after injection is common practice in the staging and surveillance of lymphoma but this procedure may not be optimal, especially not in settings where benign inflammatory lesions are of clinical concern.

In an attempt to find an alternative method for this discrimination, dual time point FDG-PET was introduced. This technique has shown itself to be a potentially promising method in FDG-PET imaging for distinguishing between malignant and benign lesions using SUV values. The reason for the different FDG uptake patterns between inflammatory and malignant lesions is unclear. Several factors may contribute to this phenomenon on a cellular basis. It has been shown that cancer cells exhibit increased numbers of glucose transporter and low level of glucose-6-phosphatase. Varying levels between different cancer cell types may explain the different FDG uptake curves. Because various cell types exhibit varying rates of FDG uptake we believe that kinetic investigation may prove to be of value in understanding different types of lymphoma and identifying how to perform precise imaging for staging and surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Planned for curative treatment

Exclusion Criteria:

* Previously treatment with chemotherapy or irradiation
* Primary CNS lymphoma
* Recurrent lymphoma
* Transformation from indolent lymphoma
* Presence of diabetes mellitus, HIV, chronic inflammatory disease or infections
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed NHL and HL
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-02 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years
  To evaluate the predictive value of PET after 60min compared to PET after 180min in terms of outcome.
Progression free survival | 3 years
  To evaluate the predictive value of PET after 60min compared to PET after 180min in terms of outcome.

SECONDARY OUTCOMES:
Overall survival | 2 years, 3 years
  To evaluate the predictive value of PET after 60min compared to PET after 180min in terms of outcome.

OTHER OUTCOMES:
To compare SUVmax with the expression of GLUT1, hexokinase, G6Pase in lymphoma cells | 1 day (After diagnostic biopsy)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Odense University Hospital, Department of hematology, Odense
  - Roskilde Hospital, Roskilde